CLINICAL TRIAL: NCT03883555
Title: High-flow Nasal Therapy for Early Management of Hypercapnic Respiratory Failure Due to Acute Cardiogenic Pulmonary Edema in the ED: a Prospective Observational Study
Brief Title: High Flow Nasal Cannula Therapy for Early Management of Acute Hypercapnic Cardiogenic Pulmonary Edema in the Emergency Department
Acronym: preopticap
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0457
Record Dates: First submitted 2019-03-06; First posted 2019-03-21 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Acute Cardiogenic Pulmonary Edema; Hypercapnic Respiratory Failure
Keywords: Acute cardiogenic pulmonary; Respiratory failure; Hypercapnia; High flow nasal oxygen; Non invasive ventilation; Emergency department
MeSH Terms: conditions — Respiratory Insufficiency; Hypercapnia; Emergencies | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Optiflow tm: High flow nasal therapy (HFNT)
  Interventions: Device: High flow nasal therapy (HFNT) : Optiflow™
- Non invasive ventilation (NIV): Non invasive ventilation (NIV)
  Interventions: Device: Non invasive ventilation (niv)

INTERVENTIONS:
Device: High flow nasal therapy (HFNT) : Optiflow™ — HFNT will be administered through a heated humidifier (Airvo 2, Fisher and Paykel healthcare) and applied through large bore binasal prongs.
  Initial gas flow rate will be set at of 60 l/min and adjusted to 40-50 l/min based on patient's tolerance. FiO2 will be adjusted to maintain an SpO2 ≥ 92%. Initial temperature will be set at 37° and reduced according to patient's tolerance
  Other Names: High flow nasal cannula; High flow nasal oxygen; Optiflow™
  Groups: Optiflow tm
Device: Non invasive ventilation (niv) — NIV will be delivered through a face mask connected to a dedicated ventilator with pressure support applied in a noninvasive ventilation mode (Monnal T75, Airliquide Medical Systems, Antony, France).
  The Pressure-support level will be adjusted to obtain an expired tidal volume of 6-8 ml/kg of predicted body weight and a respiratory rate of 25-30 b/min. PEEP (range 5-10 cm of water) and FiO2 will be adjusted to maintain an SpO2 ≥92% and to patient's comfort.
  Groups: Non invasive ventilation (NIV)

SUMMARY:
High flow nasal therapy (HFNT) has not been well evaluated for treating hypercapnia The purpose of this study is to determine whether high flow nasal therapy (HFNT) can decrease hypercapnia and improve respiratory distress parameters in Emergency Department patients with acute hypercapnic respiratory failure related to cardiogenic pulmonary edema and to compare its efficacy to that of non invasive ventilation.

DETAILED DESCRIPTION:
This is a prospective observational study conducted as a preliminary study to the randomized controlled OPTICAP trial (NCT02874339).

Prospective observational exploratory study including ED patients with a suspected diagnosis of acute hypercapnic respiratory failure related to cardiogenic pulmonary edema who require NIV according to the joint recommendations from the French society of anaesthesia and intensive care and the French society for intensive care.

Patients will receive a 1hr treatment session by either NIV or HFNT, depending on the attending ED physician expertise in using HFNT Repeat evaluation of arterial blood gases and respiratory parameters and dyspnea will be performed before and after treatment sessions according to current guidelines.

Improvement in PaCO2 and other respiratory parameters after 1hr treatment by HFNT will be analysed and compared to that of NIV.

ELIGIBILITY:
Inclusion criteria:

a suspected diagnosis of acute cardiogenic pulmonary edema presenting with any of the following criteria:

* dyspnea (orthopnea or a worsening of dyspnea according to NYHA criteria)
* respiratory rate >20 b/min
* bilateral crepitant rales at pulmonary auscultation
* pulmonary infiltrate on chest X-ray

signs of respiratory failure or any of the following clinical, laboratory or radiology signs:

* Use of accessory respiratory muscles or paradoxical abdominal movement
* Cardiomegaly (cardiothoracic ratio >0.5)
* Hypertensive crisis
* PaO2/FiO2 ≤ 300 mmHg breathing O2> 8L/min or PaO2 ≤ 63mmHg breathing room air

hypercapnia (PaCO2>45 mmHg at arterial blood gas analysis)

Exclusion criteria:

* acute exacerbation of chronic obstructive pulmonary disease or associated dyspnea from non cardiac origin
* Fever (>38,5°), sepsis or ongoing infection
* Contra-indication to NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted for acute respiratory failure secondary to acute cardiogenic lung edema with hypercapnia
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Change in PaCO2 after a 1-hour treatment session | 1 hour
  PaCO2 will be measured from standard laboratory arterial blood gas analysis performed at the end of the first 1-hour-treatment session

SECONDARY OUTCOMES:
blood gas (PaO2, pH, SaO2) | at 1 hour
  blood gas (PaO2, pH, SaO2) measured from standard laboratory arterial blood gas analysis at the end of each 1h-ventilatory support session and throughout ventilatory support
Respiratory rate | at 1 hour
  Respiratory rate, measured over 1-min as part of standard clinical assessment after each 1h ventilatory support session and throughout ventilatory support
signs of increased work of breathing | at 1 hour
  signs of increased work of breathing assessed based on patient's use of accessory respiratory muscles and paradoxical abdominal movement and measured using 5-point likert scales ranging from 1 to 5. Signs of increased work of berthing will be assessed at the end of each 1h ventilatory support sessions throughout ventilatory support
Dyspnea | at 1 hour
  Dyspnea recorded by the patient using a Modified Borg scale ranging from 0 to 10.
  Dyspnea will be measured at the end of each 1h ventilatory support sessions and throughout ventilatory support
comfort | at 1 hour
  Comfort recorded by the patient using a visual analog scale from 0 to 10. Comfort will be assessed at the end of each 1h ventilatory support sessions and throughout ventilatory support
Proportion of patients | at 1 hour
  Proportion of patients with a normalized PaCO2 (PaCO2 equal or lower than 45 mmHg),

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha Sebbane, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marjanovic N, Flacher A, Drouet L, Gouhinec AL, Said H, Vigneau JF, Chollet B, Lefebvre S, Sebbane M. High-Flow Nasal Cannula in Early Emergency Department Management of Acute Hypercapnic Respiratory Failure Due to Cardiogenic Pulmonary Edema. Respir Care. 2020 Sep;65(9):1241-1249. doi: 10.4187/respcare.07278. Epub 2020 Apr 14. PMID 32291308